CLINICAL TRIAL: NCT06740760
Title: Autism Genomics Sweden - AuGeS - Genetic Information and Guidance in Autism and Related Psychiatric Conditions Trial
Brief Title: Autism Genomics Sweden - Genetic Guidance and Information Trial
Acronym: AuGeS-GV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kristiina Tammimies, Docent (Associate Professor), Senior Researcher, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-06737-01
Record Dates: First submitted 2024-12-14; First posted 2024-12-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Autism; Autism Spectrum Disorder; ADHD - Attention Deficit Disorder With Hyperactivity; Depression Anxiety Disorder; Depression - Major Depressive Disorder; Anxiety
Keywords: genetic information; polygenic scores; rare variants; genetic counselling; genetic knowledge
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; Anxiety Disorders | interventions — Genetic Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinician led genetic information session (Active Comparator): Clinician-led structured genetic information session in person or through an online video link. Participants with genetic information available (clinically significant rare variants from exome sequencing and copy number variant analysis, and polygenic scores (autism, ADHD, depression, and anxiety), these will also be communicated as the last part of the session.
  Interventions: Behavioral: Genetic counselling
- Leaflet genetic information (Active Comparator): The participants receive a leaflet with genetic information without in-person contact
  Interventions: Behavioral: Leaflet

INTERVENTIONS:
Behavioral: Genetic counselling — Behavioral: genetic counselling
  Arms: Clinician led genetic information session
Behavioral: Leaflet — Genetic information as a form of a leaflet
  Arms: Leaflet genetic information

SUMMARY:
This observational clinical trial aims to evaluate whether providing genetic information about the origins of autism and related psychiatric disorders enhances understanding, well-being, and empowerment in adolescents and young adults with autism. The study will compare the outcomes of two groups: one receiving a 1.5-hour genetic counseling session with a clinician and the other receiving general genetic information via a leaflet. Participants will be assessed using pre- and post-intervention questionnaires, including measures of understanding of their condition (mGCOS-24) and mental health (GAD-7 and PHQ-9). The study also explores whether mental health factors like anxiety and depression influence the effectiveness of the interventions.

DETAILED DESCRIPTION:
The goal of this observational clinical study is to assess whether receiving genetic information about the origins of autism and related neuropsychiatric disorders, either at a population level or as individual information after genetic testing, can improve understanding of their condition, well-being, and empowerment in adolescents and young adults with autism spectrum condition (ASC). The main questions to answer are:

* Does a genetic counseling session improve participants' understanding of autism and its origins, well-being, and empowerment as measured by the modified Genetic Counseling Outcome Scale (mGCOS-24)?
* Is the outcome modified by mental health indicators such as anxiety and depression measures, and does the information improve these?
* We will also assess how genetic knowledge and beliefs before the genetic information session affect the main outcome of the mGCOS-24 change.

The comparison will be made between the group receiving a 1.5-hour genetic counseling session with a clinician and a group receiving general genetic information via leaflet by email to see if the genetic information session by the clinician leads to greater improvements in understanding, empowerment, and well-being.

Participants will:

* Answer basic demographic questionnaire as well as a questionnaire about genetic knowledge and beliefs
* Be randomized to receive a 1-1.5 hour genetic counseling session in person or online, or general genetic information via leaflet.
* Complete pre- and post-intervention questionnaires, including the mGCOS-24, GAD-7, and PHQ-9.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 15 - 30 years of age.
* Living in Sweden.
* Able to consent independently or with guardian consent if necessary.
* Understanding of Swedish-language questions.
* Interest in receiving genetic counselling information on autism.

Exclusion Criteria:

* Participants unwilling to complete pre- or post-intervention surveys.
* Participants unwilling to participate in either form of genetic counseling

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
modified Genetic Counselling Scale - 24 (mGCOS-24) | At enrollment (pre), 1-2 weeks after intervention (post)
  Measures changes in empowerment, understanding, and ability to use genetic information.
  Additional information: The mGCOS has been translated into Swedish based on the GCOS-validated Swedish translation.
  Change in the primary outcome will be compared between the two groups of active interventions. Subgroup analyses will be performed based on those receiving their personal genetic information vs those receiving only general population-level information.

SECONDARY OUTCOMES:
Generalised Anxiety Disorder Questionnaire (GAD-7) | Pre - Post (1-2 weeks)
  We will monitor the change in GAD-7 from pre to post.
Patient Health Questionnaire (PHQ-9) | Pre - Post (1-2 weeks)
  Evaluates changes in participants' depression symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Kristiina Tammimies, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The data dictionary will be shared openly; however, the individual-level data will be restricted to necessary clearance from the Karolinska Institutet and the Swedish Ethical Review Authority through the KI Data Repository.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: March 2025 -